CLINICAL TRIAL: NCT00822367
Title: Assessment of Glycemic Response to Commercial Nutritional Supplements in Patients With Type 2 Diabetes Mellitus
Brief Title: Blood Sugar Response to Commercial Nutritional Supplements in Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Walter Reed Army Medical Center (U.S. Federal Agency)
Responsible Party: Asha Jain, M.A., R.D., C.D.E., Walter Reed Army Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 06-10010
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Last update posted 2009-01-14 (Estimated); Status verified 2009-01

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Glucerna

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nutritional suplements (Experimental)
  Interventions: Dietary Supplement: Glucerna; Ensure; SlimFast

INTERVENTIONS:
Dietary Supplement: Glucerna; Ensure; SlimFast — Each participant will consume all three nutritional supplements randomly assigned by computer program to drink one of the three products in one week intervals. Each product will contain 50 grams of carbohydrate but differs in volume, fat, protein, and fiber composition. BG will be tested by finger sticks before (fasting) and at 15, 30, 60, 90, 120, 150 and 180 minutes after drinking the supplement. The participants will have 8 finger stick blood sugar measurements over about 3 hours on each of the 3 testing days.
  Other Names: Glucerna Weight Loss Shake;Ensure with Fiber;SlimFast Shake

SUMMARY:
The purpose of the study is to determine which of the commonly used meal supplements is the best product for patients with DM. This is important because meal supplements are becoming more popular as meal replacements in the United States. Peak blood sugar occurs about 2 hours later after a meal. Therefore, the best product would be the one that produces a smallest rise in blood sugar.

DETAILED DESCRIPTION:
The purpose of the study is to determine which of the commonly used commercial nutritional supplements are preferential for patients with Diabetes Mellitus (DM). We will compare the post-prandial blood glucose (BG) responses in response to 3 different nutritional supplements each containing 50 grams of carbohydrate in adult patients with type 2 diabetes mellitus and relate these responses to one of the two well-recognized indices of insulin sensitivity - HOMA-R and QUICKI.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-75 years
* Type-2 diabetes mellitus for over 3 months
* A1c of 7.0 - 10.0% within the past 3 months
* Controlled with diet /exercise and/or on oral anti-diabetic agents which are non-insulin secretatgogues, i.e. Metformin and/or Pioglitazone
* Able to give informed consent
* Expected to be in the DC metropolitan for the duration of the study
* Fasting blood glucose between 70 and 250 mg/dl

Exclusion Criteria:

* Patients with type 2 diabetes mellitus treated with insulin secretagogues (sulfonylurea and non-sulfonylurea), pramlintide (Symlin), GLP-1 analogs (Byetta), insulin, or alpha-glycosidase inhibitors
* A1c under 7.0% or over 10.0%
* Fasting blood glucose < 70 or > 250 mg/d
* Gastrointestinal disorders affecting digestion and absorption of nutrients such as lactose intolerance, chronic diarrhea, pancreatic insufficiency.
* Clinical history of documented gastroperesis.
* Patients on hemodialysis or peritoneal dialysis
* Pregnancy
* Inability to read and/or speak English

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2006-05; Primary Completion 2007-08 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
To determine the nutritional supplements glycemic response in patients with DM, defined as the maximum glucose excursion, area under the curve, and 2 and 3 hour BG levels fol | BG will be tested by finger sticks before (fasting) and at 15, 30, 60, 90, 120, 150 and 180 minutes after drinking the supplement.

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Vigersky, COL. MC. MD., Study Director — Walter Reed Army Medical Center